CLINICAL TRIAL: NCT00856102
Title: Efficacy of Exercise in Promotion Cognitive-psychosocial Functions in Men With Prostate Cancer Receiving Androgen Depletion Therapy
Brief Title: Exercise and Cognitive-psychosocial Functions in Men With Prostate Cancer Receiving Androgen Depletion Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: C. Ellen Lee,, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2008:318
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Control (No Intervention)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — Home-base walking program
  Arms: Exercise
Behavioral: Control — Usual care
  Arms: Control

SUMMARY:
The objective of the proposed research is to determine the efficacy of a home-based walking exercise program in promoting cognitive-psychosocial functions of men with prostate cancer receiving androgen depletion therapy (ADT). ADT is the mainstay treatment for men with advanced prostate cancer. However, ADT has a number of side effects including compromised cognitive function, depression and anxiety, which negatively impacts the quality of life of men with prostate cancer. The central question of the proposed research is to determine if exercise will have a positive impact on the quality of life of men with prostate cancer undergoing ADT.

Hypothesis:

ELIGIBILITY:
Inclusion Criteria:

* men aged 50 or older
* diagnosed with adenocarcinoma prostate cancer
* will initiate and receive continuous ADT (LHRH or combination of LHRH and anti-androgen for at least 6 months

Exclusion Criteria:

* severe cardiac disease (New York Heart Association class III or greater)
* angina
* severe osteoporosis
* uncontrolled hypertension
* orthostastic blood pressure drop > 20mm Hg
* moderate to severe aortic stenosis
* acute illness or fever
* uncontrolled atrial or ventricular dysrhythmias
* uncontrolled sinus tachycardia (> 120 beats per minute)
* uncontrolled congestive heart failure
* third-degree atrio-ventricular heart block
* active pericarditis or myocarditis
* recent embolism, thrombophlebitis
* deep vein thrombosis, resting ST displacement
* uncontrolled diabetes
* uncontrolled pain
* cognitive impairment
* history of falls due to balance impairment or lost of consciousness
* severe neuromusculoskeletal conditions that limit their ability to perform walking exercise

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cognitive-psychosocial functions | 3 and 6 months

SECONDARY OUTCOMES:
health-related quality of life | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Lee CE, Kilgour A, Lau YK. Efficacy of walking exercise in promoting cognitive-psychosocial functions in men with prostate cancer receiving androgen deprivation therapy. BMC Cancer. 2012 Jul 30;12:324. doi: 10.1186/1471-2407-12-324. PMID 22846379